CLINICAL TRIAL: NCT00004868
Title: A Phase I/II Trial of SU5416 in Patients With Recurrent High Grade Astrocytomas or Mixed Gliomas
Brief Title: SU5416 in Treating Patients With Recurrent Astrocytoma or Mixed Glioma That Has Not Responded to Radiation Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTC-9902; CDR0000067527 (Registry Identifier: PDQ (Physician Data Query)); MSKCC-01045; NCI-00-C-0173; NCT00006067 (obsolete NCT alias)
Record Dates: First submitted 2000-03-07; First posted 2003-05-23 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult meningioma; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Meningioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — Semaxinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
RATIONALE: SU5416 may stop the growth of astrocytoma or glioma by stopping blood flow to the tumor.

PURPOSE: Phase I/II trial to study the effectiveness of SU5416 in treating patients who have recurrent astrocytoma or mixed glioma that has not responded to previous radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: Phase I:

* Determine the maximum tolerated dose of SU5416 in patients with recurrent malignant glioma who are, as well as those who are not, taking enzyme-inducing antiepileptic drugs.
* Determine the toxic effects (safety profile) of this drug in this patient population.
* Characterize the pharmacokinetics of this drug in these patients.
* Develop exploratory data relative to surrogate endpoints of angiogenic activity in vivo, including functional imaging and in vitro assays of endothelial cell inhibition and serum angiogenic peptides.

Phase II:

* Determine the efficacy of SU5416, in terms of 6-month progression-free survival, in patients with recurrent high-grade glioma.
* Determine, further, the safety profile of the phase II dose of this drug in this patient population.
* Develop exploratory data relative to surrogate endpoints of angiogenic activity in vivo including functional imaging and in vitro assays of endothelial cell inhibition and serum angiogenic peptides.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to concurrent enzyme-inducing antiepileptic drugs (no vs yes).

Patients receive SU5416 IV on days 1 and 4 weekly for 4 weeks. Courses repeat every 4 weeks in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of SU5416 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD has been determined, additional patients are accrued to the phase II portion of the study. These patients receive SU5416 IV, as in the phase I portion, at the appropriate MTD established in phase I.

Patients are followed for survival.

PROJECTED ACCRUAL: At least 30 patients will be accrued for the phase I dose-escalation portion of this study within 10 months. An additional 48 patients (32 with glioblastoma multiforme and 16 with anaplastic glioma) will be accrued for the phase II portion of this study within 6-8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven supratentorial malignant primary glioma, including:

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified
  * Benign or malignant meningiomas, including brain and spinal meningiomas
* Patients with meningiomas are excluded from phase II portion of study
* Must have shown unequivocal evidence of tumor recurrence or progression by CT scan or MRI
* Must have failed prior radiotherapy
* Must have prestudy contrast MRI or contrast CT scan of brain on stable steroid dose within the past 14 days

  * Must be on stable (unchanged) dose of steroids for at least 5 days before scans
* Phase II:

  * Must have completed radiotherapy at least 2 months prior to enrollment

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* WBC at least 2,300/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL (transfusion allowed)

Hepatic:

* SGOT less than 2.5 times upper limit of normal
* Bilirubin normal
* No significant active hepatic disease

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No significant active renal disease

Cardiovascular:

* No uncompensated coronary artery disease on ECG or physical examination
* No history of myocardial infarction or severe/unstable angina within the past 6 months
* No deep venous or arterial thrombosis within the past 3 months

Pulmonary:

* No pulmonary embolism within the past 3 months

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 2 months after study
* No other serious concurrent illness
* No significant active psychiatric disease
* No diabetes mellitus with severe peripheral vascular disease
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No serious active infection
* No other concurrent disease that would obscure toxic effects or dangerously alter drug metabolism

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy (e.g., interferon) and recovered
* No concurrent immunotherapy

Chemotherapy:

* Phase I:

  * No more than 2 prior chemotherapy regimens for recurrent disease
* Phase II:

  * No more than 1 prior chemotherapy regimen for recurrent disease
* At least 2 weeks since prior vincristine
* At least 6 weeks since prior nitrosoureas
* At least 3 weeks since prior procarbazine
* Recovered from prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 3 weeks since prior endocrine therapy (e.g., tamoxifen) and recovered

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* Recovered from prior surgery
* Recent prior resection of recurrent or progressive tumor allowed

Other:

* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03-24 (Actual); Primary Completion 2004-09-15 (Actual); Study Completion 2005-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Fine, MD, Study Chair — NCI - Neuro-Oncology Branch
Locations (12):
- United States (12):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Neuro-Oncology Branch, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin